CLINICAL TRIAL: NCT00757315
Title: Prospective, Controlled Study of the Efficacy of NdYag for Acne Keloidalis Nuchae
Brief Title: NdYag Laser for Acne Keloidalis Nuchae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5244
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Acne Keloidalis Nuchae; NdYag Laser; AKN; Acne Keloidalis; AK; Dermatitis Papillaris Capillitii; Folliculitis Keloidalis Nuchae; Sycosis Nuchae; Acne Keloid; Keloidal Folliculitis; Lichen Keloidalis Nuchae; Folliculitis Nuchae Scleroticans; Sycosis Framboesiformis
Keywords: acne keloidalis nuchae; NdYag laser; AKN; acne keloidalis; AK; dermatitis papillaris capillitii; folliculitis keloidalis nuchae; sycosis nuchae; acne keloid; keloidal folliculitis; lichen keloidalis nuchae; folliculitis nuchae scleroticans; sycosis framboesiformis
MeSH Terms: conditions — Acne Keloid | interventions — Adrenal Cortex Hormones; Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: NdYag Laser(hair removal laser) plus topical corticosteroid
- 2 (Active Comparator)
  Interventions: Drug: Topical corticosteroid alone

INTERVENTIONS:
Device: NdYag Laser(hair removal laser) plus topical corticosteroid — NdYag laser and topical corticosteroid are applied to one half of the scalp.
  Other Names: triamcinolone
  Arms: 1
Drug: Topical corticosteroid alone — topical corticosteroid alone is applied to one half of the scalp
  Other Names: Triamcinolone
  Arms: 2

SUMMARY:
Acne Keloidalis Nuchae (AKN) is a long standing hair follicle disease with bumps and scars on the skin of the back of the head and neck. The purpose of this new study is to determine how well a hair removal laser (NdYag Laser) works in treating AKN.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, the subject must:

  1. Be at least 18 years old
  2. Be otherwise healthy
  3. Have a diagnosis of AKN with at least 10 papules/pustules and/or a non-keloidal plaque > 7 cm2 in area.

Exclusion Criteria:

* Subject must not:

  1. Have AKN with a keloidal plaque >3 cm in length
  2. Be using any other medications or undergoing any other procedures for the treatment of AKN
  3. Have used any topical medications or undergone any procedures for the treatments of AKN within two weeks of study enrollment
  4. Have used any oral medications for AKN within 4 weeks of study enrollment:
  5. Have serious, uncontrolled medical conditions
  6. Be pregnant at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
reduction in severity of AKN as measured by a novel AKN severity scoring system which incorporates number of lesions, size of lesions, type of lesions and associated inflammation. | 6 months

SECONDARY OUTCOMES:
Treatment tolerability as measured by 0 to 10 pain scale | 6 months
treatment safety | 6 months
  This will be assessed by the frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Health Systems Dermatology Department
Locations (1):
- Henry Ford Medical Center, New Center One, Detroit, Michigan, United States

REFERENCES:
- [Background] Battle EF Jr, Hobbs LM. Laser-assisted hair removal for darker skin types. Dermatol Ther. 2004;17(2):177-83. doi: 10.1111/j.1396-0296.2004.04018.x. PMID 15113285
- [Background] Shah GK. Efficacy of diode laser for treating acne keloidalis nuchae. Indian J Dermatol Venereol Leprol. 2005 Jan-Feb;71(1):31-4. doi: 10.4103/0378-6323.13783. PMID 16394358